CLINICAL TRIAL: NCT06329011
Title: Combining Transcranial Direct Current Stimulation With Intermittent Oral to Esophageal Tube for Stroke-related Dysphagia Management: Double Blind Randomized Controlled Study
Brief Title: Combining Transcranial Direct Current Stimulation With Intermittent Oral to Esophageal Tube for Stroke-related Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDC+IOE
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive rehabilitation+Intermittent Oro-esophageal Tube+Transcranial stimulation (Experimental): The patients are randomly assigned to either the experimental group or the placebo group. All patients receive routine rehabilitation therapy and swallowing rehabilitation training, along with enteral nutrition support using Intermittent Oro-esophageal Tube. In addition to these interventions, patients in the experimental group receive transcranial direct current stimulation, while the instruments used for patients in the placebo group only illuminate an indicator light without any actual effect.
  Interventions: Behavioral: Comprehensive rehabilitation therapy; Device: Intermittent Oro-esophageal Tube Feeding; Device: Transcranial direct current stimulation
- Comprehensive rehabilitation+Intermittent Oro-esophageal Tube (Placebo Comparator): The patients are randomly assigned to either the experimental group or the placebo group. All patients receive routine rehabilitation therapy and swallowing rehabilitation training, along with enteral nutrition support using Intermittent Oro-esophageal Tube. In addition to these interventions, patients in the experimental group receive transcranial direct current stimulation, while the instruments used for patients in the placebo group only illuminate an indicator light without any actual effect.
  Interventions: Behavioral: Comprehensive rehabilitation therapy; Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: Placebo Transcranial direct current stimulation

INTERVENTIONS:
Behavioral: Comprehensive rehabilitation therapy — Including： Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
Device: Intermittent Oro-esophageal Tube Feeding — All patients are given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure: Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
Device: Transcranial direct current stimulation — In this study, transcranial direct current stimulation is performed using a battery-powered constant current stimulator. This device delivers the current through two electrodes immersed in saline solution. Specifically, a 50mm*50mm anodal electrode pad is placed at the center of the healthy side swallowing sensory-motor cortex of the patient. According to the positioning method of the international 10-20 electrode system, the swallowing sensory-motor cortex of the left brain is located at the midpoint between C3 and T3, while that of the right brain is located at the midpoint between C4 and T4. The cathode is placed on the opposite shoulder, using a current of 1mA, once a day, for 20 minutes each time, and 5 days a week. The instruments used for placebo patients will not have any actual effect.
  Arms: Comprehensive rehabilitation+Intermittent Oro-esophageal Tube+Transcranial stimulation
Behavioral: Placebo Transcranial direct current stimulation — The Transcranial direct current stimulation will be performed without being turned on.
  Arms: Comprehensive rehabilitation+Intermittent Oro-esophageal Tube

SUMMARY:
The study is a double-blind randomized controlled trial, lasting for 15 days for each participant. Patients with post-stroke dysphagia who receive treatment at the Rehabilitation Department are selected as the study subjects. The patients are randomly assigned to either the experimental group or the placebo group. All patients receive routine rehabilitation therapy and swallowing rehabilitation training, along with enteral nutrition support using Intermittent Oro-esophageal Tube. In addition to these interventions, patients in the experimental group receive transcranial direct current stimulation, while the instruments used for patients in the placebo group only illuminate an indicator light without any actual effect.

DETAILED DESCRIPTION:
Transcranial direct current stimulation is currently very popular. The study is a double-blind randomized controlled trial, lasting for 15 days for each participant. Patients with post-stroke dysphagia who receive treatment at the Rehabilitation Department are selected as the study subjects. The patients are randomly assigned to either the experimental group or the placebo group. All patients receive routine rehabilitation therapy and swallowing rehabilitation training, along with enteral nutrition support using Intermittent Oro-esophageal Tube. In addition to these interventions, patients in the experimental group receive transcranial direct current stimulation, while the instruments used for patients in the placebo group only illuminate an indicator light without any actual effect.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for ischemic stroke confirmed by MRI or CT;
* Age > 18 years;
* First-time stroke;
* Swallowing disorder confirmed by swallowing contrast study or flexible endoscopic evaluation of swallowing;
* Requires enteral nutrition support;
* Stable vital signs, no severe cognitive impairment or aphasia, able to cooperate with treatment;
* Transferred to the rehabilitation department within fifteen days of onset;
* Stable vital signs.

Exclusion Criteria:

* Presence of contraindications for invasive oral endoscopy;
* Concurrent presence of other neurodegenerative diseases that may cause swallowing disorders, such as neurodegenerative diseases;
* Concurrent presence of other neurological disorders;
* Tracheostomized patients;
* Concurrent liver, kidney failure, tumor, or hematological disorders;
* Pregnancy;
* Presence of contraindications for transcranial direct current stimulation, such as epilepsy, cerebral edema;
* Recent use of centrally acting drugs that interfere with the effects of transcranial direct current stimulation, such as carbamazepine, phenytoin, valproic acid, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | day 1 and day 15
  Penetration-Aspiration Scale is used to measure swallowing safety, which is also the primary outcome of this study. Before and after treatment, patients are required to undergo a swallow study to complete the assessment. This scale evaluates the patient's swallowing function level and aspiration risk by assessing leakage and aspiration during the patient's swallowing process. The scale ranges between level 1 and level 8, with higher levels indicating poorer swallowing function and lower swallowing safety (worse outcomes).

SECONDARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 15
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.
Swallowing Quality of Life Questionnaire | day 1 and day 15
  The Swallowing Quality of Life Questionnaire (SWAL-QOL) is used to evaluate the impact of swallowing function on patients' quality of life. The questionnaire consists of 44 questions related to swallowing function and quality of life. Each question is answered using a 5-point rating scale. In this study, the final score is converted into a percentage. The higher scores indicate the better quality of life.
Patient Health Questionnaire-9 | day 1 and day 15
  To assess the patients' depression levels, a questionnaire is used. The questionnaire consists of 9 questions related to depressive symptoms, and each question is answered using a 4-point rating scale. The total score ranges from 0 to 27, with higher scores indicating a greater tendency towards depression.
Body weight | day 1 and day 15
  Body weight measurement of the infants was conducted by the same nurse according to the relevant standards.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Study Chair — Site Coordinator of United Medical Group located in Miami